CLINICAL TRIAL: NCT06541938
Title: A Feasibility Study to Use a Handheld, In-Home Breath Test Device to Measure H2 and CH4 Production from Carbohydrate Fermentation and Its Correlation with Persistent Symptoms in Inflammatory Bowel Disease Patients in Remission
Brief Title: AIRE-2 Device for Study of Breath Analysis in IBD
Acronym: AIRE-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, David Armstrong, Professor, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 17342
Record Dates: First submitted 2024-07-10; First posted 2024-08-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: We have 2 groups (IBD patients & healthy controls) so 30 per group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case - Inflammatory Bowel Disease (Experimental): Patients with IBD, under clinical remission since more than 3 months, having at least one symptom
  Interventions: Dietary Supplement: low FODMAP diet; Dietary Supplement: Lactose Sachet; Dietary Supplement: Fructose Sachet; Dietary Supplement: Sorbitol Sachet; Dietary Supplement: Inulin Sachet; Device: AIRE-2 Portable breath analyzer
- Control - Healthy household member (Active Comparator): Family member of IBD patients who lives in the same house, shares similar diet and has no active GI disease or symptom
  Interventions: Dietary Supplement: low FODMAP diet; Dietary Supplement: Lactose Sachet; Dietary Supplement: Fructose Sachet; Dietary Supplement: Sorbitol Sachet; Dietary Supplement: Inulin Sachet; Device: AIRE-2 Portable breath analyzer

INTERVENTIONS:
Dietary Supplement: low FODMAP diet — You consume low FODMAP diet for 24 hours before taking the FODMAP challenge
Dietary Supplement: Lactose Sachet — You will engage in a 4-week study to document responses to 4 Fermentable Carbohydrates(FCHOs): Lactose(25g), Fructose(25g), Sorbitol(10g), and Inulin(10g). Each FCHO, dissolved in 250ml of lukewarm water, is taken after a 24-hour low FODMAP diet to clear residual FCHOs. Exhaled H2 and CH4 are measured before and 60 minutes after the first and last meal of the low FODMAP period. Each morning, after a baseline breath test, you will consume one FCHO challenge and record breath tests for three hours at 15-minute intervals. Following each challenge, there is a 6-day washout period with your typical diet. This 24-hour low FODMAP diet, FCHO challenge, and washout cycle is repeated until all FCHOs are tested. The order of FCHO challenges is randomized and consistent among all, who remain blinded to the order to minimize confounding factors.
  25g sachet having lactose roughly equal to amount of lactose present in 1 large glass of milk
Dietary Supplement: Fructose Sachet — You will engage in a 4-week study to document responses to 4 Fermentable Carbohydrates(FCHOs): Lactose(25g), Fructose(25g), Sorbitol(10g), and Inulin(10g). Each FCHO, dissolved in 250ml of lukewarm water, is taken after a 24-hour low FODMAP diet to clear residual FCHOs. Exhaled H2 and CH4 are measured before and 60 minutes after the first and last meal of the low FODMAP period. Each morning, after a baseline breath test, you consume one FCHO challenge and record breath tests for three hours at 15-minute intervals. Following each challenge, there is a 6-day washout period with your typical diet. This 24-hour low FODMAP diet, FCHO challenge, and washout cycle is repeated until all FCHOs are tested. The order of FCHO challenges is randomized and consistent among all, who remain blinded to the order to minimize confounding factors.
  25g sachet having fructose roughly equal to the amount of fructose present in 2 large apples
Dietary Supplement: Sorbitol Sachet — You will engage in a 4-week study to document responses to 4 Fermentable Carbohydrates(FCHOs): Lactose(25g), Fructose(25g), Sorbitol(10g), and Inulin(10g). Each FCHO, dissolved in 250ml of lukewarm water, is taken after a 24-hour low FODMAP diet to clear residual FCHOs. Exhaled H2 and CH4 are measured before and 60 minutes after the first and last meal of the low FODMAP period. Each morning, after a baseline breath test, you consume one FCHO challenge and record breath tests for three hours at 15-minute intervals. Following each challenge, there is a 6-day washout period with your typical diet. This 24-hour low FODMAP diet, FCHO challenge, and washout cycle is repeated until all FCHOs are tested. The order of FCHO challenges is randomized and consistent among all, who remain blinded to the order to minimize confounding factors.
  10g sachet of sorbitol is roughly equal to the amount of sorbitol present in 3 pears or 1 prune
Dietary Supplement: Inulin Sachet — You will engage in a 4-week study to document responses to 4 Fermentable Carbohydrates(FCHOs): Lactose(25g), Fructose(25g), Sorbitol(10g), and Inulin(10g). Each FCHO, dissolved in 250ml of lukewarm water, is taken after a 24-hour low FODMAP diet to clear residual FCHOs. Exhaled H2 and CH4 are measured before and 60 minutes after the first and last meal of the low FODMAP period. Each morning, after a baseline breath test, you consume one FCHO challenge and record breath tests for three hours at 15-minute intervals. Following each challenge, there is a 6-day washout period with your typical diet. This 24-hour low FODMAP diet, FCHO challenge, and washout cycle is repeated until all FCHOs are tested. The order of FCHO challenges is randomized and consistent among all, who remain blinded to the order to minimize confounding factors.
  A 10g sachet of inulin is roughly equal to the amount of inulin present in 1 head of garlic
Device: AIRE-2 Portable breath analyzer — The AIRE-2 breath analyzer will capture hydrogen and methane at baseline and after every fodmap challenge

SUMMARY:
The goal of this Prospective single-blinded intervention feasibility study is the utilization of the AIRE-2 device and FoodMarble app to elucidate the interplay among diet, symptoms, and microbial fermentable features in IBD patients with persistent intestinal symptoms and their household controls.

AIRE-2 captures exhaled hydrogen and methane and FoodMarble app records breath levels, symptoms and dietary intake.

The main questions it aims to answer are:

1. To assess the feasibility of using the AIRE-2 device, FoodMarble mobile app in a cohort of IBD patients and their household controls to collect data on diet, symptoms and exhaled H2 and CH4 levels. 2.
2. To assess the feasibility of using FoodMarble's FODMAP discovery kit protocol in a cohort of IBD patients and their household controls.
3. To collect preliminary data on the relation between diet, symptoms, and exhaled H2 and CH4 levels measured by the AIRE-2 device and FoodMarble app in a cohort of IBD patients and their household controls.
4. To explore the correlation between the fecal microbiome sequencing profile with exhaled H2 and CH4 levels, diet and symptoms in a cohort of IBD patients and their household controls.

You will:

1. Record regular diet in the FoodMarble app and collect baseline stool samples
2. You will then take a low FODMAP diet for 24 hours every week and record the diet and symptoms. After the diet, you will take the FODMAP challenge of Lactose, Fructose, Sorbitol and Inulin (one every week) using Sachets provided by FoodMarble company, record exhaled breath levels, symptoms and collect stool. This process will take 4 weeks.
3. Visit clinic to submit stool samples

DETAILED DESCRIPTION:
Study Design Type:

Prospective single-blinded intervention feasibility study

Methodology/Study Design:

A cohort of IBD patients and their healthy household controls will be recruited for this study. You will be instructed to use a handheld breathalyzer device, AIRE-2, to measure exhaled H2 and CH4 gas production, and its smartphone app, FoodMarble, will be used to log your diet and symptoms for a period of 5 weeks, as follows:

AIRE-2 will be used before and after two meals each day - the first meal and the last meal of the day. You will breathe into the AIRE-2 device before eating to obtain the baseline value. After the meal, you will breathe into the AIRE-2 60 minutes postprandially. The exhaled H2 and CH4 measurements will be automatically logged into the FoodMarble app, which is connected via Bluetooth. You will log your food intake and symptoms in FoodMarble. Symptoms scores will be recorded at the same time that the AIRE- 2 device is being used - 60 minutes postprandial. You will be asked not to drink alcohol during the meals that will be recorded, as this will skew the device results. You will be informed that you can consume alcoholic drinks after doing the postprandial breath test.

Study procedure:

1. Study Enrolment and Familiarization Period: At visit 1, you will be trained to use the AIRE-2 device which McMaster has purchased from the FoodMarble company and will be provided to you. You will also be trained to use the FoodMarble app. The FoodMarble company is the owner of the AIRE-2 device which is being used in the present study, the company wouldn't have access to resulting data other than publication. Demographics, medical history, disease activity, Gastrointestinal symptom rating scale (GSRS), Bristol stool type, medications, supplements, perceived food intolerances and general dietary patterns will be recorded at baseline. We shall assist you in inputting some GI and extra-intestinal symptoms (headache, foggy mind, numbness of joints, joint pain, fainting, oral lesions, dermatitis) manually in the FoodMarble app from the GSRS symptom questionnaire as all symptoms are not mentioned in the app and there is a provision to edit the symptom list. After visit 1, you will have 3 days to use the device and app in order to become familiar with its use and report any challenges and difficulties to us in visit 2 (online via McMaster Zoom). At the end of the familiarization period, you are expected to be comfortable using the AIRE-2 device and the FoodMarble app. No data reported during this period will be used for the purpose of analysis or outcomes evaluation.
2. Baseline Period: This period starts after the familiarization week and runs for one week, representing the beginning of the data tracking collection. During the baseline period, you will eat your normal, typical diet, while collecting your breath test, food and symptoms as described above. The baseline period serves to capture the natural fluctuations of breath H2 and CH4 of each individual and to explore the correlations with diet and symptoms. You will be instructed to take the breath test before and 60 minutes after two major meals, every day. You will also collect the baseline stool sample and drop it off at the study location during visit 3, at the end of this period. You will be handed the low FODMAP diet chart which will be required in discovery period.
3. Discovery Period: This period starts after the baseline period and runs for four weeks. During this period, you will document your responses to challenges with four specific FCHOs)- Lactose, Fructose, Sorbitol, and Inulin ("Food Intolerance Kit", FoodMarble Inc, Dublin, Ireland). The quantities of each FCHO challenge are as follows: lactose and fructose sachets, 25g each. A sachet of lactose roughly equal to amount of lactose present in 1 large glass of milk. A sachet of fructose is roughly equal to amount of fructose present in 2 large apples. Sorbitol and inulin sachets contain 10g each. A sachet of sorbitol is roughly equal to the amount of sorbitol present in 3 pears or 1 prune. A sachet of inulin is roughly equal to the amount of inulin present in 1 head of garlic. Each sachet has to be dissolved in 250 ml of lukewarm water. Before each challenge, you will follow a low FODMAP diet for 24h to facilitate clearance of any FCHOs from the intestine. You will be guided by a registered dietitian (RD) regarding an appropriate low FCHO diet, supported by the FoodMarble app, which provides a large database of low FODMAP meals and recipes. You will log all meals during the 24h low FCHO period using the FoodMarble app. The meals will be analyzed by the RD and scored, on a 4-point scale (poor, moderate, good, excellent) for adherence to the low FCHO diet. Exhaled H2 and CH4 will be measured before and 60 min after the first and last meal during this period, as usual. After the 24h low FCHO diet, you will consume one FCHO challenge in the morning (after the baseline breath test) and take the postprandial breath test 60 min later. You will be required to record the breath test for 3 hours after every 15 minutes as per the protocol of the kit. You will then collect the first stool sample after the challenge and submit it to us in visit 4. Symptoms and meals will continue to be logged in the FoodMarble app. You will also be instructed to fill in a validated questionnaire to assess symptoms before and after the FCHO challenge (Adult Carbohydrate Perception Questionnaire). This questionnaire will be given to you in paper form. A 6-day washout period will be implemented in between the FCHO challenges. During the washout period, you will follow your typical diet. The 24h low Fodmap day, FCHO challenge, 6-day washout cycle and submission of stool samples (visit 4-7) will be repeated until all 4 FCHO challenges have been completed. The order of the FCHO challenges will be randomized and will be kept constant between all of you to minimize potential co-founding factors related to the order of the intervention. However, you will be blinded to the order.
4. End of the study: At the end of the discovery period, you will answer a feedback survey to report their experience using AIRE-2 and FoodMarble.

ELIGIBILITY:
Inclusion criteria (IBD):

* Age 18-75 years old, confirmed diagnosis of IBD (UC or CD)
* Under clinical remission for at least 3 months
* Report having one or more IBS-like symptom (abdominal pain, altered bowel habit, flatulence, abdominal distension etc)
* Own a smartphone with Bluetooth capability
* Fluent in English.
* Able to understand the instructions to use smartphone apps
* Able to provide informed consent

Exclusion criteria (IBD):

* Use of antibiotics 1 month before enrolment
* Active IBD (disease activity score, fecal calprotectin, CRP)
* History of bowel resection
* Presence of a stoma
* Pregnancy
* Type 1 diabetes or insulin-dependent Type 2 diabetes
* Currently being treated for eating disorder, schizophrenia, psychosis or other acute mental disorder

A total of 30 adult IBD patients (18-75 years old), 15 ulcerative colitis (UC) and 15 Crohn's disease (CD) patients, will be recruited at the Digestive Diseases Clinic, McMaster University, Hamilton, Ontario.

Controls: A total of 30 non-IBD volunteers from the same household as the recruited IBD patients who do not have any IBS-like symptom will be recruited as controls.

Inclusion criteria:

* Age 18-75 years old, IBS-negative (Rome IV negative)
* Living in the same household as IBD patients, sharing a similar diet
* Asymptomatic
* Own a smartphone with Bluetooth capability
* Fluent in English.
* Able to understand the instructions to use smartphone apps
* Able to provide informed consent

Exclusion criteria:

* Diagnosed with IBD or other Gastrointestinal disorder
* Use of antibiotics 1 month before enrolment
* Pregnancy
* Type 1 diabetes or insulin-dependent Type 2 diabetes
* Currently being treated for eating disorder, schizophrenia, psychosis or other acute mental disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proof of data collection/Adherence to the protocol | 40 months
  For each data set, we will divide the number of logged data divided by the total data expected to be logged. For example, the number of breath tests using AIRE-2 logged by the participant / total expected. This will also apply to the diet log. The results will be expressed in %.

SECONDARY OUTCOMES:
Comparison of positive breath between IBD and non-IBD patients | 40 months
  average of # >3 breath test score / total group #
Prevalence of positive score with symptoms between IBD and non-IBD patients | 40 months
  # of events when >3 breath test score match with symptomatic event / total positive test events
Correlation of positive breath tests with severity of symptoms | 40 months
  using person correlation coefficient
Correlation of breath scores with food reported as being intolerant by the patients | 40 months
  matching between reported dietary triggers at baseline and positive breath test
Microbiome taxa | 40 months
  We will explore the correlation between the presence of microbiome genera with the exhaled H2 and CH4 scores. The microbiome profile will be done by 16S rRNA sequencing of fecal samples.
Relative abundance of predicted microbial metabolic pathways | 40 months
  Microbial metabolic pathways will be predicted using PICRUSt and correlated with dietary intake and breath test results

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada